CLINICAL TRIAL: NCT04341506
Title: Evaluating Non-contact ECG Sensor System for Early Detection of COVID19
Brief Title: Non-contact ECG Sensor System for COVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Andrew Gostine, MD, Doctor, Northwestern Medicine
Other Study IDs: 20-0407
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: COVID-19; ECG; Arrhythmia
MeSH Terms: conditions — COVID-19; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Participant ECG: The study has one arm, I.e., we will collect daily ECGs in 100 participants and track their ECG over three months. We will then compare ECGs pre and post COVID-19 diagnosis in any participant diagnosed with COVID-19 to assess for any early ECG changes that may aid with diagnosing.
  Interventions: Device: Non-contact ECG

INTERVENTIONS:
Device: Non-contact ECG — A non-contact ECG will be used to detect a patient cardiac electrical activity.

SUMMARY:
The purpose of this study is two-fold. First we would like to confirm that non-contact ECG provides equivalency to current contact methods of obtaining ECG data. Second we would like to investigate whether non-contact ECG can detect ECG changes prior to the onset symptoms from COVID19.

ELIGIBILITY:
Inclusion Criteria:

* Any employee of Lake Forrest Memorial Hospital presenting to work
* Age greater than 18 years-old

Exclusion Criteria:

* Age less than 18 years-old
* Non-employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 employees of Lake Forrest Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
ECG changes associated with COVID-19 | 3 months
  Assess different ECG changes in participants diagnosed with COVID-10

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No